CLINICAL TRIAL: NCT04888689
Title: Holter of Movement in Patients with Multiple Sclerosis. Acti-SEP Study: Controlled Environment.
Brief Title: Holter of Movement in Patients with Multiple Sclerosis in Controlled Environment.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laurent Servais (Other)
Collaborators: SYSNAV (Industry); Centre Hospitalier Régional de la Citadelle (Other)
Responsible Party: Sponsor-Investigator, Laurent Servais, Principal investigator, Centre Hospitalier Universitaire de Liege
Organization: Centre Hospitalier Universitaire de Liege (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ActiSEP. Part 1.
Record Dates: First submitted 2021-03-11; First posted 2021-05-17 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Multiple Sclerosis
Keywords: Actimyo; Accelerometry; Motion laboratory
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: all patients undergo clinical evaluation while wearing Actimyo device to assess their gait.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MS patients (Experimental): Ambulant patients with multiple sclerosis
  Interventions: Device: Actimyo°; Device: IMU

INTERVENTIONS:
Device: Actimyo° — Actimyo° is an innovative device intended to be used in a home-based environment. It is composed of two watch-like sensors, each containing a magneto-inertial sensors that record the linear acceleration, the angular velocity, the magnetic field of the movement in all directions.The two watches can be worn as wristwatch or placed near the ankle.
Device: IMU — IMU is a portable system of miniaturized inertial sensors for objective, instrumental, ambulatory, and validated analysis of normal and pathological human gait. Each miniaturized inertial sensor (2 cm × 0.7 cm × 0.5 cm) includes a triaxial accelerometer and a triaxial gyroscope.
  These four inertial sensors are connected to a box by wires and are numbered 1 to 4. They must be attached - using adhesive tapes - on the participant's shoes.

SUMMARY:
ActiSEP is a multicentric academic study. Ambulant patients with multiple sclerosis may be included on a voluntary basis. We plan to include a group of approximately 20 patients with MS.

This study include a unique evaluation in the laboratory of analysis of human movement. A set of tasks will be performed by patients wearing of two magneto-inertial sensors.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed MS diagnosis,
* Over 18 years old,
* Ambulant patients,
* Signed informed consent,
* No clinical and / or radiological relapse within 3 months.

Exclusion Criteria:

* Patients with excessive cognitive disorders, limiting the understanding of task or with apparent communication difficulties hindering data collection.
* Any other previous or present pathology having an impact on motor function.
* Recent surgery or trauma (less than 6 months) in the upper or lower limbs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-02-04 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
95th centile of stride velocity | One day
  95th centile of stride velocity obtained with magneto-inertial sensors and a motion capture device (meter/second).
50th centile of stride velocity | One day
  50th centile of stride velocity obtained with magneto-inertial sensors and a motion capture device (meter/second).
95th centile of stride length | One day
  95th centile of stride length obtained with magneto-inertial sensors and a motion capture device (meter).
50th centile of stride length | One day
  50th centile of stride length obtained with magneto-inertial sensors and a motion capture device (meter).
Stance phase time | One day
  Stance time over full stride time for each foot obtained with magneto-inertial sensors and a motion capture device (percentage).

CONTACTS AND LOCATIONS:
Overall Officials: Margaux Poleur, MD, Principal Investigator — CHR Citadelle-CHU liège
Locations (1):
- Centre Hospitalier Régional de la Citadelle, Liège, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No